CLINICAL TRIAL: NCT04044755
Title: Investigating the Effect of Using Myopia Prediction Algorithm on Myopia Children's Eye Refraction in China: a Multi-center Randomized Control Trial
Brief Title: Investigating the Effect of Using Myopia Prediction Algorithm on Myopia Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CCPMOH2019-China-3
Record Dates: First submitted 2019-08-02; First posted 2019-08-05 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors involved in data management and analysis will be blinded to the group assignment. The study participants, the investigators responsible for randomization will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using myopia prediction algorithm (Experimental): After examination of visual acuity, eye refraction and biometrics, the examination results are shown to the children. Meanwhile, myopia prediction algorithm will be used to predict SER at 3 years.
  Interventions: Other: Myopia prediction algorithm
- Not using myopia prediction algorithm (No Intervention): After examination of visual acuity, eye refraction and biometrics, the examination results are shown to the children.

INTERVENTIONS:
Other: Myopia prediction algorithm — Candidate predictors mainly includes age at examination, SER, and annual progression rate. Using these predictors, the algorithm will be used to predict SER at 3 years.
  Arms: Using myopia prediction algorithm

SUMMARY:
In this study, the investigators aim to perform a prospective, randomized controlled study to compare the myopia development between myopia children using myopia prediction algorithm and myopia children without using myopia prediction algorithm

DETAILED DESCRIPTION:
We propose to enroll myopia children aged 8-10 in China. Children will be given examinations of visual acuity, eye refraction and biometrics, and be assigned to two groups: participants in group A use myopia prediction algorithm to predict myopia development, while in Group B, the participants do not use myopia prediction algorithm to predict myopia development. The visual acuity, eye refraction and biometrics will be investigated over the one-year follow-up period, aiming at comparison of actual myopia development between the two groups

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-10
* Has the record of eye refraction examined in the past year, SER<-0.5D
* Current BCVA≥0.8, SER<-0.5D, Astigmatism less than 1.50 D, anisometropia less than 1.50 D
* Written informed consents provided

Exclusion Criteria:

* Definitive diagnosis of other diseases except for refractive error
* Previous eye surgery
* Previous usage of orthokeratology lenses and atropine
* Unwilling to participate in this trial

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2138 (Estimated)
Dates: Start 2019-08-03 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of SER development of at least -0.5 dioptres (D) | up to 1 year
  SER: spherical equivalent refraction, sphere + ½ 360 cylinder; SER development of at least -0.5 dioptres: SER2 - SER1≤-0.5D; SER1: SER at baseline; SER2: SER up to 1 year

SECONDARY OUTCOMES:
Incidence of SER development of at least -1.0 dioptres (D) | Up to 2 year
  SER: spherical equivalent refraction, sphere + ½ 360 cylinder; SER development of at least -1.0 dioptres: SER2 - SER1≤-0.5D; SER1: SER at baseline; SER2: SER up to 2 year
Changes in SER \ and AL | Up to 1 year
  Changes in SER \ and AL will be calculated; AL: axial length
Changes in SER \ and AL | Up to 2 year
  Changes in SER \ and AL will be calculated; AL: axial length
Changes in proportion of children using atropine | Up to 1 year
  Changes in proportion of children using atropine will be calculated
Changes in proportion of children using atropine | Up to 2 year
  Changes in proportion of children using atropine will be calculated
Changes in proportion of children using orthokeratology lenses | Up to 1 year
  Changes in proportion of children using orthokeratology lenses will be calculated
Changes in proportion of children using orthokeratology lenses | Up to 2 year
  Changes in proportion of children using orthokeratology lenses will be calculated
Changes in proportion of children using spectacles | Up to 1 year
  Changes in proportion of children using spectacles will be calculated
Changes in proportion of children using spectacles | Up to 2 year
  Changes in proportion of children using spectacles will be calculated
Changes in child's average outdoor activity time per day | Up to 1 year
  Changes in child's average outdoor activity time per day will be calculated
Changes in child's average outdoor activity time per day | Up to 2 year
  Changes in child's average outdoor activity time per day will be calculated
Changes in child's average screen time per day | Up to 1 year
  Changes in child's average screen time per day will be calculated
Changes in child's average screen time per day | Up to 2 year
  Changes in child's average screen time per day will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Centre, Guangzhou, Guangdong, China